CLINICAL TRIAL: NCT01175681
Title: Effect of Remote Ischemia Preconditioning on Myocardial Injury in Patients Undergoing Heart Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangzhou First People's Hospital (Other)
Responsible Party: Jing-song Ou/ professor, The First Affiliated Hospital, Sun Yat-sen University.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ischemia
Record Dates: First submitted 2010-08-03; First posted 2010-08-05 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Heart Valve Diseases
Keywords: rheumatic heart disease; degenerated heart valve disease; heart valve prolapse
MeSH Terms: conditions — Heart Valve Diseases; Rheumatic Heart Disease; Heart Valve Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment (Experimental): remote ischaemic preconditioning
  Interventions: Procedure: remote ischaemic preconditioning
- untreated (No Intervention): control

INTERVENTIONS:
Procedure: remote ischaemic preconditioning — Remote ischaemic preconditioning consisted of three 5-min cycles of right upper arm ischaemia, which was induced by an automated cuff -inflator placed on the right upper arm and inflated to 200 mm Hg, with an intervening 5 min of reperfusion during which the cuff was deflated. There was a 5- to 10-min interval between completion of the remote ischaemic preconditioning protocol and initiation of bypass.Control patients had a deflated cuff placed on the right upper arm for 30 min.
  Arms: treatment

SUMMARY:
Remote ischaemic preconditioning has shown its cardiac protective effect during heart surgery including coronary artery bypass graft surgery, congenital heart disease and aneurysm. However, no data was reported on heart valve disease surgery. Rheumatic heart disease is one of the major heart diseases requiring surgery in China. Thus, the investigators chose heart valve disease as a focus to see whether remote ischaemic preconditioning also has cardiac protective effect during heart valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* All heart valve diseases needing heart valve surgery.

Exclusion Criteria:

* All four limbs existed ischemic condition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-12; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
plasma troponin I level | with 7 days after surgery
  The investigators will measure the plasma troponin I level in several time points before and after surgery in each patient.

SECONDARY OUTCOMES:
serum creatinine | within 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jing-song Ou, MD,PhD, Principal Investigator — The Frist Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Derived] Xie JJ, Liao XL, Chen WG, Huang DD, Chang FJ, Chen W, Luo ZL, Wang ZP, Ou JS. Remote ischaemic preconditioning reduces myocardial injury in patients undergoing heart valve surgery: randomised controlled trial. Heart. 2012 Mar;98(5):384-8. doi: 10.1136/heartjnl-2011-300860. Epub 2011 Nov 22. PMID 22107759
- See also: Pubmed — http://www.ncbi.nlm.nih.gov